CLINICAL TRIAL: NCT01360476
Title: Adjunct Vitamin D Therapy as a Means to Reduce the Disparity in Subclinical Target Organ Cardiac Damage Among Vulnerable Hypertensive Patients
Brief Title: Vitamin D Therapy to Reduce Cardiac Damage Among Vulnerable Hypertensive Patients
Acronym: AdDReaCH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wayne State University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Phillip D. Levy, Associate Director of Clinical Research, Wayne State University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1R01MD005849-01A1 (NIH)
Record Dates: First submitted 2011-05-19; First posted 2011-05-25 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Hypertension; Left Ventricular Hypertrophy
Keywords: hypertension; left ventricular hypertrophy; Vitamin D; African-Americans
MeSH Terms: conditions — Hypertension; Hypertrophy, Left Ventricular | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D (Active Comparator)
  Interventions: Dietary Supplement: cholecalciferol (Vitamin D)
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol (Vitamin D) — 50,000 UI, chewable wafer every 2 weeks for 52 weeks (27 total doses)
  Arms: Vitamin D
Dietary Supplement: Placebo — chewable wafer every 2 weeks for 52 weeks (27 total doses)
  Arms: placebo

SUMMARY:
This project seeks to reduce the disparity in hypertensive heart disease which exists for African-Americans who have poorly controlled hypertension (HTN), also known as blood pressure (BP). The investigators are targeting a highly vulnerable, often neglected subject population which stands to benefit tremendously from better BP control and a corresponding decrease in heart damage. HTN occurs early in life and more often in African-Americans, reducing both quality and quantity of life. Inner-city African-Americans with HTN utilize the emergency department (ED) for chronic BP management. Like cardiovascular disease, vitamin D deficiency disproportionately affects African-Americans. Vitamin D is thought to play an important role in cardiovascular health. Vitamin D replacement in those who are deficient has been thought to reduce the cardiovascular disease, especially if initiated early before irreversible damage has occurred, but this has yet to be tested in a prospective clinical trial. Accordingly, this proposal was designed to investigate the relationship between vitamin D and cardiac damage (as identified on cardiac magnetic resonance imaging) in a cohort of African-American, vitamin D deficient hypertensive patients without prior history of heart disease.

The primary objective of this proposal is to evaluate the efficacy of vitamin D therapy in vitamin D deficient African-Americans with HTN. Vitamin D is an inexpensive treatment, which, if shown to be effective could improve the existing approach to a widely accessible, cost-effective option.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with known HTN
* African-American race (self reported)
* Repeat SBP ≥ 160 mmHg within 1 hour of arrival
* Age 30-74 years
* Asymptomatic state (class I as defined by Goldman Specific Activity Scale)

Exclusion Criteria:

* Dyspnea (exertional, rest or nocturnal) or chest pain as a primary or secondary chief complaint
* Prior history of HF, coronary artery disease, myocardial infarction, cardiomyopathy (any), valvular heart disease (any) or renal failure with current, previous, or planned future dialysis
* Acute illness or injury which necessitates hospital admission
* Acute alcohol or cocaine intoxication or history of chronic alcohol (determined using the CAGE screening questions) or cocaine (self-reported) abuse
* Acute or decompensated psychiatric disorder or any underlying psychiatric disorder or cognitive deficit which precludes effective on-going communication or ability to follow-up as required
* Cancer (other than skin), HIV, or any other medical condition that might limit life expectancy
* Hepatitis or liver enzyme (ALT, AST) elevations > 1.5x normal
* Planned move > 50 miles in the next 9 months
* History of kidney stones
* GFR <30
* Serum calcium > 10.5 mg/dl or known history of hypercalcemia
* History of or known primary hyperparathyroidism
* Sarcoidosis or other granulomatous disease
* Pregnant or planning to become pregnant
* Allergy or known hypersensitivity to gadolinium contrast
* Severe claustrophobia

Ages: 30 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 354 (Actual)
Dates: Start 2011-08; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in left ventricular hypertrophy at 1 year | baseline, 16weeks, 52weeks
  Cardiac MRI will be used to assess this change.

CONTACTS AND LOCATIONS:
Overall Officials: Phillip D Levy, MD, Principal Investigator — Wayne State University
Locations (1):
- Detroit Receiving Hospital, Detroit, Michigan, United States